CLINICAL TRIAL: NCT00198705
Title: Community Based Interventions to Reduce Neonatal Mortality in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Shimantik, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Abdullah Baqui, Professor, International Health and Director, International Center for Maternal and Newborn Health, Johns Hopkins Bloomberg School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H.22.00.12.06.BX
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

INTERVENTIONS:
Behavioral: Improved management of severe neonatal infections

SUMMARY:
This project delivers, promotes and facilitates services related to pregnancy, delivery and newborn care.

DETAILED DESCRIPTION:
The Project entitled "Community-Based Intervention to Reduce Neonatal Mortality in Bangladesh", also known as Projahnmo - I (Project to Advance the Health of Newborns and Mothers), is a partnership project of the Johns Hopkins Bloomberg School of Public Health (JHSPH), USA, with a number of Bangladeshi organizations including: a) the Ministry of Health and Family Welfare (MOHFW) of the Government of Bangladesh (GoB), b) the Centre for Health and Population Research (ICDDRB), c) Save the Children/USA, Bangladesh Field Office (SC/BFO), d) Shimantik, a Bangladeshi NGO, e) BRAC/Bangladesh, f) Dhaka Shishu Hospital and g) the Institute of Child and Mother Health (ICMH). The project is funded through four mechanisms: 1) USAID Global funding to cover expenses of JHSPH to design and to provide technical assistance in the implementation and evaluation of the various components of the project, 2) SNL/SC funding to JHSPH to sub-contract the Bangladeshi institutions listed above to support implementation of the intervention component of the project, 3) USAID/Bangladesh funding to ICDDRB to cover the cost of implementation of the research and evaluation component of the project, 4) the Bangladeshi government's contribution in-terms of staff time, supplies, and facilities. This partnership between multiple research institutions and donors brings diverse, rich and unique experiences and expertise. It ensures the relevance of the project and increases the likelihood of scaling up and sustaining the intervention.

The goals of Projahnmo I are to: (a) introduce two models of delivering improved maternal and newborn care in rural Bangladesh; (b) measure each model's impact on neonatal mortality and other relevant indicators; (c) assess the cost effectiveness and feasibility of the two models.

The project includes two intervention arms with two different service delivery models, home care (HC) and clinic care (CC). Community health workers (CHWs) and community mobilizers (CMs) deliver the Birth and Newborn Care Preparedness (BNCP) package, which includes counseling during the antenatal period, delivery care, care of the baby during delivery, postnatal care, and continued counseling and education during the neonatal period. Service provision also includes making referral for sick newborns and playing the role of facilitator for behavior change in the households and communities. The strategic approaches used also include pregnancy surveillance and community-level mobilization of specific target groups, such as pregnant women, senior female family members, husbands and other targeted local advocacy meetings. In both arms, community-based meetings conducted by CMs focus on facilitating involvement of the mothers and other family members in the decision-making process and making them aware of the importance of proper antenatal care, delivery care, postpartum care, and newborn care. In the HC model, counseling is conducted at home with pregnant women and their families by CHWs. In the CC arm, women receive these messages through community meetings by CMs and during antenatal check-up (ANC) visits by governmental primary health workers and paramedics. In CC arms, CMs identify community change agents to assist in creating awareness and promoting behavior change. In addition, traditional birth attendants (TBAs), who commonly attend home deliveries in the study communities, have been oriented on newborn health.

ELIGIBILITY:
Inclusion Criteria:

* participants consenting for the home-based care model area
* participants who consent for household adequacy survey
* participants who consent from clinic care model area

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10670 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality rate

SECONDARY OUTCOMES:
Neonatal colonization with antibiotic-resistant bacteria
Cost of providing the intervention services per neonate

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Baqui, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Baqui AH, Ahmed S, El Arifeen S, Darmstadt GL, Rosecrans AM, Mannan I, Rahman SM, Begum N, Mahmud AB, Seraji HR, Williams EK, Winch PJ, Santosham M, Black RE; Projahnmo 1 Study Group. Effect of timing of first postnatal care home visit on neonatal mortality in Bangladesh: a observational cohort study. BMJ. 2009 Aug 14;339:b2826. doi: 10.1136/bmj.b2826. PMID 19684100
- [Derived] Baqui AH, El-Arifeen S, Darmstadt GL, Ahmed S, Williams EK, Seraji HR, Mannan I, Rahman SM, Shah R, Saha SK, Syed U, Winch PJ, Lefevre A, Santosham M, Black RE; Projahnmo Study Group. Effect of community-based newborn-care intervention package implemented through two service-delivery strategies in Sylhet district, Bangladesh: a cluster-randomised controlled trial. Lancet. 2008 Jun 7;371(9628):1936-44. doi: 10.1016/S0140-6736(08)60835-1. PMID 18539225